CLINICAL TRIAL: NCT05552703
Title: Traumatic Extradural Hematoma in Paediatric Age Group
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Salah, Principal Investigator,, Assiut University
Other Study IDs: EDH in paediatric
Record Dates: First submitted 2021-11-17; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Extradural Hematoma
Keywords: paediatrics
MeSH Terms: conditions — Hematoma, Epidural, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: surgical evacuation of extradural hematoma — evacuation of extradural hematoma by craniotomy

SUMMARY:
The aim of this study is to assess the clinical and radiological characteristics of children with traumatic extradural hematoma and factors affecting the initial neurological status and outcome.

DETAILED DESCRIPTION:
Extradural hematoma (EDH) represents 2.7-4% of traumatic brain injury .EDH is a potentially lethal condition which is easily cured if diagnosed early .EDH is less frequent in pediatric age group than in adults. The mean age of pediatric patients harboring EDH is between 6 and 10 years and it is rare among infants under the age of 12 months. EDH in children differs significantly from adults in terms of mode of injury, prognostic factors, and outcome. EDH in children may follow a trivial trauma and the course is more insidious and associated skull fractures is less frequent and these factors make it difficult to diagnose and often challenging to manage. The reported rate of mortality from EDH in children is varying from 0% and 17%, The criteria for choosing the surgical evacuation Vs. conservative management in pediatric age group still ill-defined this is what encouraged the investigators to carry this study to present our experience in the management of EDH in children aged less than 18 years.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients with traumatic extradural hematoma presenting at our institute and managed surgically.

Exclusion Criteria:

* Patients aged more than 18 years old.
* patients with other traumatic brain injuries like: acute subdural hematoma, intra-cerebral hematoma and subarachnoid hemorrhage.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with traumatic extradural hematoma presenting at our institute and managed surgically.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
glascow outcome scale | immediately after the intervention/procedure/surgery
  The Glasgow Outcome Scale (GOS) categorizes the outcomes of patients after traumatic brain injury, as follows
  1. Persistent vegetative state: Minimal responsiveness
  2. Severe disability: Conscious but disabled; dependent on others for daily support
  3. Moderate disability: Disabled but independent; can work in sheltered setting
  4. Good recovery: Resumption of normal life despite minor deficits

SECONDARY OUTCOMES:
mortality | immediately after the intervention/procedure/surgery, through study completion, an average of 1 year
  patients who died after surgery
morbidity | immediately after the intervention/procedure/surgery, through study completion, an average of 1 year
  patients with disability after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://link.springer.com/article/10.1007/BF01808613